CLINICAL TRIAL: NCT01427036
Title: Impact Sur le Saignement Per et Post opératoire de 2 stratégies d'ostéosynthèse Des Fractures du Massif trochantérien du Sujet > 65 Ans : Essai randomisé Comparant le système MISS et le système PHS
Brief Title: On the Impact of Bleeding on Two Strategies Osteosynthesis of Trochanteric Fractures
Acronym: MISSvsPHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRI/09/PR/MISSvsPHS; ID RCB 2009-A00713-54 (Other: AFSSaPS)
Record Dates: First submitted 2011-05-31; First posted 2011-09-01 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2018-10

CONDITIONS: Other Reconstructive Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MISS surgery group (Experimental): hip screw MISS® (Minimally Invasive Screw System) : minimally invasive approach
  Interventions: Procedure: MISS
- PHS surgery group (Active Comparator): PHS® hip screw design for standard approach
  Interventions: Procedure: PHS

INTERVENTIONS:
Procedure: MISS — Installation of the patient in the operating room (same technique for MISS and PHS) operated supine on a fracture table, a fluoroscope (C Arm) authorizing a control AP and lateral.
  Reduction of the fracture before incision (same technique for MISS and PHS): it is essential for minimally invasive surgery and inclusion in the study. One checked on the AP and the lateral view the absence of a fracture gap greater than the thickness of the the cortical.
  skin incision 6 to 8 cm in the axis of the proximal femur, beginning a little above trochanteric crest in, then incised longitudinally extensive externe1 cm under the sub trochanteric crest, on a length of 3 cm. Passage of the raspatory along thefemoral shaft under the muscle on the entire length of the plate.
  Other Names: dynamic hip screw
  Arms: MISS surgery group
Procedure: PHS — Installation of the patient in the operating room (same technique for MISS and PHS) operated supine on a fracture table, a fluoroscope (C Arm) authorizing a control AP and lateral.
  Reduction of the fracture before incision (same technique for MISS and PHS): it is essential for minimally invasive surgery and inclusion in the study. One checked on the AP and the lateral view the absence of a fracture gap greater than the thickness of the the cortical.
  Surgical approach for PHS : Longitudinal external starting on trochanteric crest, long 15-20 cm depending on morphotype of the patient. Incision of the fascia latta like a " L " detaching the vastus lateralis to expose the external surface of the femur on the length of the plate.
  Other Names: Pertrochanteric Hip Screw
  Arms: PHS surgery group

SUMMARY:
Fractures of the trochanter in the elderly have a terrible prognosis both vital and functional. It is certainly possible to reduce the medical and economic impact of this disease by reducing surgical trauma, by means of minimally invasive osteosynthesis material adapted to this approach. This minimally invasive approach should, however, guarantee a result at least equal to the standard approach. The goal is to have a technique, easily to transmit, using a percutaneous approach, but which may be converted to conventional surgery in case of difficulty, and with implants appropriate for trochanteric fractures.

With this in mind, the dynamic hip screw MISS® (Minimally Invasive Screw System) was developed and has already demonstrated its effectiveness in terms of anatomical results. It is as effective than the PHS® hip screw design for standard approach. The two implants have the same plate and screw and differ only by the system for fixing the screw on the plate to allow minimal invasive approach.

DETAILED DESCRIPTION:
Fractures of the trochanter in the elderly have a terrible prognosis both vital and functional. It is certainly possible to reduce the medical and economic impact of this disease by reducing surgical trauma, by means of minimally invasive osteosynthesis material adapted to this approach. This minimally invasive approach should, however, guarantee a result at least equal to the standard approach. The goal is to have a technique, easily to transmit, using a percutaneous approach, but which may be converted to conventional surgery in case of difficulty, and with implants appropriate for trochanteric fractures.

With this in mind, the dynamic hip screw MISS® (Minimally Invasive Screw System) was developed and has already demonstrated its effectiveness in terms of anatomical results. It is as effective than the PHS® hip screw design for standard approach. The two implants have the same plate and screw and differ only by the system for fixing the screw on the plate to allow minimal invasive approach.

The main objective of the study is to show that the use of dynamic hip screw MISS is associated with lower morbidity (in terms of bleeding) in comparison with the material PHS standard (Pertrochanteric Hip Screw) implanted by standard approach.

The secondary objectives are :

* Check the quality of reduction and stability of osteosynthesis with the MISS are equivalent to those of the PHS.
* Assessing the economic impact on the duration of use of operating rooms and the length of hospitalization

The study is a randomized trial with multicenter parallel group with collection of blinded endpoint : PROBE Study (Prospective Randomized Blinded Endpoint), comparing two techniques : minimally invasive approach versus standard approach, Apart from the incision, and the system fixing the screw to the plate, all other periods of the operation will be identical. Operation is done on table fracture with X-rays control with C arm. Associated therapies will be identical in both groups and follow the protocols of the department.

Number of patients : 54 in each group = 108 patients Duration of the research Duration of the inclusion period: 21 months Duration of participation for each patient: three months Total duration of the study: 24 months

Expected effects :

For patients: intervention better supported, postoperative more simple, shortened length of stay and faster rehabilitation.

For the hospital: intervention shorter and simpler, lower occupation time of block, decreased average length of stay.

For society: reduced cost of care of these patients by society

ELIGIBILITY:
Inclusion Criteria:

Age greater than 65. Patient with a fracture of the trochanter, isolated fractures or other trauma may be increased blood loss.

Establishment of a screw-on plate hip had not had previous intervention Having signed an informed consent Member or beneficiary of a social security system Patient with the criteria for inclusion and pre- Reduced fracture on a fracture table before any incision.

Exclusion Criteria:

Delay between the onset of fracture and intervention than 7 days Polytrauma patient and "polyfracturé" Hip already made or with a degenerative, inflammatory, infectious or known or suspected tumor History of contralateral hip fracture within 12 months Impossible to reduce the fracture on a fracture table before incision History of pathology of coagulation known Proven history of allergy to LMWH

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-06; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
perioperative blood loss which is assessed between day 0 and day 5 by the following formula: | day 5
  Primary outcome measure :
  It is defined by the perioperative blood loss which is assessed between day 0 and day 5 by the following formula:
  PBL = BVT x ΔHt + 150 x PRBC where: PBL = Perioperative Blood Loss (mL) between day 0 and day 5 BVT = Blood Volume Theorical (mL) = 70ml/kg humans, 65ml/kg in non-obese women ΔHt = (preoperative hematocrit at D0) - (Hct on day 5 postoperative) 150 (ml) = average volume of unit of Packed Red Blood Cells PRBC = number of Packed Red Blood Cells administered to the patient

SECONDARY OUTCOMES:
Clinical Criteria and Radiographic criteria | 3 months
  secondary outcome measure
  Clinical Criteria:
  * Duration of hospitalization
  * Onset of complications not attributable to implant during hospitalization (thrombo-embolic. ..).
  * Intra-and postoperative complication related to the implant (fracture implant, migration of implant removal).
  * Length of the incision
  * Duration of intervention (incision to closure)
  * Rates of surgical site infection
  * Need for reoperation Radiographic criteria
  * Reduction of the fracture on X-Rays (AP and latéral)
  * Position of implants
  * Consolidation
  * Secondary displacement

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROSSET, Pr, Principal Investigator — Service d'Orthopédie II - CHRU de TOURS
Locations (2):
- France (2):
  - CHU, Rennes
  - UH Tours CHRU Trousseau, Tours

REFERENCES:
- [Result] Besnard M, Leger J, Babusiaux D, Marty F, Ropars M, Rosset P, Le Nail LR. Comparison of bleeding during trochanteric fracture fixation with mini-invasive or conventional side plate fixation: A randomized controlled trial. Orthop Traumatol Surg Res. 2023 Nov;109(7):103661. doi: 10.1016/j.otsr.2023.103661. Epub 2023 Jul 18. PMID 37474020